CLINICAL TRIAL: NCT06552702
Title: Race and Socioeconomic Position: Examining Common Social Pathways to Disease Risk
Status: Completed | Type: Observational
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: 21044507
Record Dates: First submitted 2023-06-29; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Healthy Aging
Keywords: socioeconomic status; race; stress; social relationships; ambulatory blood pressure

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community sample: Black Americans (8 high SEP, 8 low SEP) and White Americans (8 high SEP, 8 low SEP) between the ages of 35 and 70
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — There is no intervention.

SUMMARY:
Black Americans and those of lower socioeconomic position (SEP) are at higher risk for multiple diseases of aging and shorter lifespans, but the psychophysiological mechanisms that may account for these effects are not clear. The overarching objective of this pilot grant is to improve our understanding of the proximal social exposures and subsequent psychobiological processes that contribute to racial and socioeconomic health disparities. Precisely understanding what these mutable social and psychological mechanisms are is necessary in order to identify intervention targets at the level of the individual.

DETAILED DESCRIPTION:
Black Americans and those of lower socioeconomic position (SEP) are at higher risk for multiple diseases of aging and shorter lifespans. Though these disparities are well-documented, the mechanisms that may account for them are still poorly understood. Low income or Black race do not, themselves, cause individuals to become sick. Instead, the social context and exposures associated with these personal attributes give rise to differential risk (1-3). Black race and lower SEP are overlapping in the United States and race and SEP may share common social exposures that contribute to disease risk because both Blacks and individuals of lower SEP are socially marginalized (e.g., devalued, pushed to the lower margins of society) and thus exposed to more stress associated with lower hierarchical rank (4). However, no studies to our knowledge have been designed to examine whether day-to-day social exposures common across race and SEP may contribute to higher overall disease burden in these groups. In this project, investigators examine whether daily social interaction patterns help to explain how race and SEP may be linked with well-established psychobiological pathways to disease (affect, behavior, and physiology). With respect to each of these pathways, investigators examine the extent to which within-person changes in social processes may be associated with effects that mirror (and thus could explain) between-group differences. For example, interactions in which one experiences a higher degree of disrespect may be associated with momentary changes in affect, behavior, and physiology that confer disease risk. Examination of these within-person processes allows for stronger causal inference and is directly relevant to the development of individual-level interventions (e.g., targeting cognitive, behavioral, and affective processes). These findings can directly inform individual and group interventions for stress reduction in health disparity populations.

ELIGIBILITY:
Inclusion Criteria:

- Black American or White American between the ages of 35 and 70.

Exclusion Criteria:

* Conditions that require immediate treatment (e.g., Stage 2 hypertension; resting blood pressure > 160/100 mmHg)
* Excessive alcohol consumption (> 5 portions, > 3 times per week)
* Frequent illicit drug use
* Schizophrenia or bipolar disorder
* Permanent neurological deficit
* Shift work
* Current pregnancy

Ages: 35 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recruitment will target Black Americans (8 high SEP, 8 low SEP) and White Americans (8 high SEP, 8 low SEP) between the ages of 35 and 70. Low SEP will be defined as a score of 1 to 3 on the MacArthur (ladder) scale of subjective social status (range 1-10), and high SEP as a score of 8-10 on the same scale.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Ambulatory Systolic Blood Pressure | during four days of ambulatory monitoring
  Mean
Ambulatory Diastolic Blood Pressure | during four days of ambulatory monitoring
  Mean

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Cundiff, Principal Investigator — University of Alabama at Birmingham; Karlene Ball, Study Director — University of Alabama at Birmingham
Locations (1):
- University of AL Psychology Department, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Data will also be presented at international scientific meetings regularly attended by the PI (e.g., American Psychosomatic Society, Society for Behavioral Medicine) and shared at both national and regional RCMAR conferences. Preliminary findings from this proposed study will be used to apply for NIH R-series funding to conduct a larger study.

REFERENCES:
- [Background] Jones CP. Levels of racism: a theoretic framework and a gardener's tale. Am J Public Health. 2000 Aug;90(8):1212-5. doi: 10.2105/ajph.90.8.1212. PMID 10936998
- [Background] Bailey ZD, Krieger N, Agenor M, Graves J, Linos N, Bassett MT. Structural racism and health inequities in the USA: evidence and interventions. Lancet. 2017 Apr 8;389(10077):1453-1463. doi: 10.1016/S0140-6736(17)30569-X. PMID 28402827
- [Background] Krieger N, Chen JT, Waterman PD, Rehkopf DH, Subramanian SV. Painting a truer picture of US socioeconomic and racial/ethnic health inequalities: the Public Health Disparities Geocoding Project. Am J Public Health. 2005 Feb;95(2):312-23. doi: 10.2105/AJPH.2003.032482. PMID 15671470
- [Background] Williams DR, Mohammed SA. Racism and Health I: Pathways and Scientific Evidence. Am Behav Sci. 2013 Aug 1;57(8):10.1177/0002764213487340. doi: 10.1177/0002764213487340. PMID 24347666